CLINICAL TRIAL: NCT01686828
Title: Androgen-mediated Pathways in the Regulation of Insulin Sensitivity in Men
Brief Title: T-IR- Study to Understand the Effects of Testosterone and Estrogen on the Body's Response to the Hormone Insulin
Acronym: T-IR
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Katya Rubinow, Assistant Professor, Division of Metabolism, Endocrinology and Nutrition, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00002641
Record Dates: First submitted 2012-09-12; First posted 2012-09-18 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-04

CONDITIONS: Insulin Resistance; Type 2 Diabetes Mellitus; Obesity; Androgen Deficiency; Metabolic Disease
Keywords: insulin; androgens; insulin resistance; testosterone; estradiol; obesity
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2; Obesity; Metabolic Diseases | interventions — acyline; Testosterone; Gels; Letrozole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Acyline & placebo gel & placebo pill (Experimental): Acyline (300mcg/kg) + placebo transdermal gel + placebo pill daily
  Interventions: Drug: Acyline; Drug: Placebo gel (for Testosterone 1.62% gel); Drug: Placebo pill (for Letrozole)
- Acyline & Testosterone 1.25g & placebo pill (Experimental): Acyline (300mcg/kg) + Testosterone gel (1.25g) daily + placebo pill daily
  Interventions: Drug: Acyline; Drug: Testosterone 1.62% gel; Drug: Placebo pill (for Letrozole)
- Acyline & Testosterone 5g & placebo pill (Experimental): Acyline (300mcg/kg) + Testosterone gel (5g) daily + placebo pill daily
  Interventions: Drug: Acyline; Drug: Testosterone 1.62% gel; Drug: Placebo pill (for Letrozole)
- Acyline & Testosterone & Letrozole (Experimental): Acyline (300mcg/kg) + Testosterone gel (5g) daily + letrozole (5mg) daily
  Interventions: Drug: Acyline; Drug: Testosterone 1.62% gel; Drug: Letrozole

INTERVENTIONS:
Drug: Acyline — 300 mcg/mL administered subcutaneously (at Day 0, Week 2)
Drug: Testosterone 1.62% gel — Transdermal Testosterone Gel (either 1.25g or 5g/d) for 4 weeks
  Other Names: Androgel
  Arms: Acyline & Testosterone & Letrozole; Acyline & Testosterone 1.25g & placebo pill; Acyline & Testosterone 5g & placebo pill
Drug: Letrozole — Letrozole oral aromatase inhibitor 5mg daily for 4 weeks
  Other Names: Femara
  Arms: Acyline & Testosterone & Letrozole
Drug: Placebo gel (for Testosterone 1.62% gel) — placebo gel manufactured to mimic Testosterone 1.62% gel
  Arms: Acyline & placebo gel & placebo pill
Drug: Placebo pill (for Letrozole) — Oral placebo aromatase inhibitor to mimic Letrozole 5mg/d
  Arms: Acyline & Testosterone 1.25g & placebo pill; Acyline & Testosterone 5g & placebo pill; Acyline & placebo gel & placebo pill

SUMMARY:
The purpose of this research study is to understand the effects of testosterone and estrogen on the body's response to the hormone insulin.

DETAILED DESCRIPTION:
The investigators will examine the effects of testosterone on insulin sensitivity and body composition in men. This study may lend greater insight into the increased risk of diabetes evident in men with low circulating levels of testosterone. Three drugs will be used in this study: acyline, given by injection; testosterone (T) gel that is applied to the skin; and letrozole, which is an oral drug that blocks the conversion of androgens (male hormones) to estrogens (female hormones). Acyline inhibits the production of luteinizing hormone (LH) and follicle stimulating hormone (FSH). When acyline stops the production of these hormones, it blocks the signal from the brain that stimulates the testicles to make testosterone. Adding testosterone to acyline will restore physiologic levels of testosterone in some study participants. One group of men will receive T gel with letrozole, an aromatase inhibitor; these men will have normal levels of testosterone but low levels of estrogen in the blood. This design will enable determination of the respective metabolic effects of testosterone and estrogen.

ELIGIBILITY:
Inclusion Criteria:

* Prostate-specific antigen (PSA) ≤ 3 ng/mL
* Age 25-55 years
* Ability to understand the study, study procedures and provide informed consent
* Serum total T > 300 ng/dL
* Normal reproductive history and exam
* International Prostate Symptom Score (IPSS) < 11

Exclusion Criteria:

* A history of prostate cancer including suspicious digital rectal exam (DRE) or history of highgrade prostatic intraepithelial neoplasia (PIN) on prostate biopsy
* Invasive therapy for benign prostatic hyperplasia (BPH) in the past
* History of acute urinary retention in the previous 3 months
* Current or recent past use of androgenic or anti-androgenic drugs, steroids or drugs which interfere with steroid metabolism (within the last 3 months)
* Current use of statins or glucocorticoids
* Severe systemic illness (renal, liver, cardiac, lung disease, cancer, diabetes mellitus) or skin disease
* A history of or current breast cancer
* Known, untreated obstructive sleep apnea
* Hematocrit > 50 or < 34
* Hypersensitivity to any of the drugs used in the study
* History of a bleeding disorder or anticoagulation
* Participation in any other drug study within past 90 days
* History of drug or alcohol abuse within the last 12 months
* Weight > 280 lbs. or BMI ≥ 33
* Desire for fertility in the next 6 months or current pregnant partner
* Sperm concentration <14 million/ml
* Significant, uncontrolled hypertension (BP >160/100 mmHg); subjects with well-controlled BP on medical therapy will be eligible to participate

Ages: 25 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William J Bremner, MD, PhD, Study Chair — University of Washington; Stephanie T Page, MD, PhD, Study Director — University of Washington; Katya Rubinow, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Flegal KM. Excess deaths associated with obesity: cause and effect. Int J Obes (Lond). 2006 Aug;30(8):1171-2. doi: 10.1038/sj.ijo.0803313. No abstract available. PMID 16871273
- [Background] Araujo AB, O'Donnell AB, Brambilla DJ, Simpson WB, Longcope C, Matsumoto AM, McKinlay JB. Prevalence and incidence of androgen deficiency in middle-aged and older men: estimates from the Massachusetts Male Aging Study. J Clin Endocrinol Metab. 2004 Dec;89(12):5920-6. doi: 10.1210/jc.2003-031719. PMID 15579737
- [Background] Yeap BB, Chubb SA, Hyde Z, Jamrozik K, Hankey GJ, Flicker L, Norman PE. Lower serum testosterone is independently associated with insulin resistance in non-diabetic older men: the Health In Men Study. Eur J Endocrinol. 2009 Oct;161(4):591-8. doi: 10.1530/EJE-09-0348. Epub 2009 Aug 6. PMID 19661128
- [Background] Muller M, Grobbee DE, den Tonkelaar I, Lamberts SW, van der Schouw YT. Endogenous sex hormones and metabolic syndrome in aging men. J Clin Endocrinol Metab. 2005 May;90(5):2618-23. doi: 10.1210/jc.2004-1158. Epub 2005 Feb 1. PMID 15687322
- [Background] Li C, Ford ES, Li B, Giles WH, Liu S. Association of testosterone and sex hormone-binding globulin with metabolic syndrome and insulin resistance in men. Diabetes Care. 2010 Jul;33(7):1618-24. doi: 10.2337/dc09-1788. Epub 2010 Apr 5. PMID 20368409
- [Background] Smith MR, Lee H, Fallon MA, Nathan DM. Adipocytokines, obesity, and insulin resistance during combined androgen blockade for prostate cancer. Urology. 2008 Feb;71(2):318-22. doi: 10.1016/j.urology.2007.08.035. PMID 18308111
- [Background] Smith MR, Lee H, Nathan DM. Insulin sensitivity during combined androgen blockade for prostate cancer. J Clin Endocrinol Metab. 2006 Apr;91(4):1305-8. doi: 10.1210/jc.2005-2507. Epub 2006 Jan 24. PMID 16434464
- [Background] Mauras N, Hayes V, Welch S, Rini A, Helgeson K, Dokler M, Veldhuis JD, Urban RJ. Testosterone deficiency in young men: marked alterations in whole body protein kinetics, strength, and adiposity. J Clin Endocrinol Metab. 1998 Jun;83(6):1886-92. doi: 10.1210/jcem.83.6.4892. PMID 9626114
- [Background] Yialamas MA, Dwyer AA, Hanley E, Lee H, Pitteloud N, Hayes FJ. Acute sex steroid withdrawal reduces insulin sensitivity in healthy men with idiopathic hypogonadotropic hypogonadism. J Clin Endocrinol Metab. 2007 Nov;92(11):4254-9. doi: 10.1210/jc.2007-0454. Epub 2007 Aug 28. PMID 17726076
- [Background] Klimcakova E, Roussel B, Kovacova Z, Kovacikova M, Siklova-Vitkova M, Combes M, Hejnova J, Decaunes P, Maoret JJ, Vedral T, Viguerie N, Bourlier V, Bouloumie A, Stich V, Langin D. Macrophage gene expression is related to obesity and the metabolic syndrome in human subcutaneous fat as well as in visceral fat. Diabetologia. 2011 Apr;54(4):876-87. doi: 10.1007/s00125-010-2014-3. Epub 2011 Jan 26. PMID 21267541
- [Background] Odegaard JI, Chawla A. Mechanisms of macrophage activation in obesity-induced insulin resistance. Nat Clin Pract Endocrinol Metab. 2008 Nov;4(11):619-26. doi: 10.1038/ncpendmet0976. Epub 2008 Oct 7. PMID 18838972
- [Background] Rubinow KB, Snyder CN, Amory JK, Hoofnagle AN, Page ST. Acute testosterone deprivation reduces insulin sensitivity in men. Clin Endocrinol (Oxf). 2012 Feb;76(2):281-8. doi: 10.1111/j.1365-2265.2011.04189.x. PMID 21797916
- [Background] Ortega Martinez de Victoria E, Xu X, Koska J, Francisco AM, Scalise M, Ferrante AW Jr, Krakoff J. Macrophage content in subcutaneous adipose tissue: associations with adiposity, age, inflammatory markers, and whole-body insulin action in healthy Pima Indians. Diabetes. 2009 Feb;58(2):385-93. doi: 10.2337/db08-0536. Epub 2008 Nov 13. PMID 19008342
- [Background] Weisberg SP, McCann D, Desai M, Rosenbaum M, Leibel RL, Ferrante AW Jr. Obesity is associated with macrophage accumulation in adipose tissue. J Clin Invest. 2003 Dec;112(12):1796-808. doi: 10.1172/JCI19246. PMID 14679176
- [Background] Xu HZ, Li Y, Zhao YF. [Diagnosis and treatment of osteopathic parathyroid adenoma]. Zhongguo Xiu Fu Chong Jian Wai Ke Za Zhi. 2003 Nov;17(6):446-9. Chinese. PMID 14663938
- [Background] Lumeng CN, DelProposto JB, Westcott DJ, Saltiel AR. Phenotypic switching of adipose tissue macrophages with obesity is generated by spatiotemporal differences in macrophage subtypes. Diabetes. 2008 Dec;57(12):3239-46. doi: 10.2337/db08-0872. Epub 2008 Oct 1. PMID 18829989
- [Background] Rull A, Camps J, Alonso-Villaverde C, Joven J. Insulin resistance, inflammation, and obesity: role of monocyte chemoattractant protein-1 (or CCL2) in the regulation of metabolism. Mediators Inflamm. 2010;2010:326580. doi: 10.1155/2010/326580. Epub 2010 Sep 23. PMID 20936118
- [Background] Bastard JP, Maachi M, Lagathu C, Kim MJ, Caron M, Vidal H, Capeau J, Feve B. Recent advances in the relationship between obesity, inflammation, and insulin resistance. Eur Cytokine Netw. 2006 Mar;17(1):4-12. PMID 16613757
- [Background] Chazenbalk G, Bertolotto C, Heneidi S, Jumabay M, Trivax B, Aronowitz J, Yoshimura K, Simmons CF, Dumesic DA, Azziz R. Novel pathway of adipogenesis through cross-talk between adipose tissue macrophages, adipose stem cells and adipocytes: evidence of cell plasticity. PLoS One. 2011 Mar 31;6(3):e17834. doi: 10.1371/journal.pone.0017834. PMID 21483855
- [Background] Gilliver SC. Sex steroids as inflammatory regulators. J Steroid Biochem Mol Biol. 2010 May 31;120(2-3):105-15. doi: 10.1016/j.jsbmb.2009.12.015. Epub 2010 Jan 4. PMID 20045727
- [Background] Cunningham M, Gilkeson G. Estrogen receptors in immunity and autoimmunity. Clin Rev Allergy Immunol. 2011 Feb;40(1):66-73. doi: 10.1007/s12016-010-8203-5. PMID 20352526
- [Background] Bouman A, Moes H, Heineman MJ, de Leij LF, Faas MM. The immune response during the luteal phase of the ovarian cycle: increasing sensitivity of human monocytes to endotoxin. Fertil Steril. 2001 Sep;76(3):555-9. doi: 10.1016/s0015-0282(01)01971-9. PMID 11532481
- [Background] Lai JJ, Lai KP, Chuang KH, Chang P, Yu IC, Lin WJ, Chang C. Monocyte/macrophage androgen receptor suppresses cutaneous wound healing in mice by enhancing local TNF-alpha expression. J Clin Invest. 2009 Dec;119(12):3739-51. doi: 10.1172/JCI39335. Epub 2009 Nov 9. PMID 19907077
- [Background] Hildebrand F, Thobe BM, Hubbard WJ, Choudhry MA, Pape HC, Chaudry IH. Effects of 17beta-estradiol and flutamide on splenic macrophages and splenocytes after trauma-hemorrhage. Cytokine. 2006 Nov;36(3-4):107-14. doi: 10.1016/j.cyto.2006.11.002. Epub 2007 Jan 4. PMID 17207634
- [Background] Qiu Y, Yanase T, Hu H, Tanaka T, Nishi Y, Liu M, Sueishi K, Sawamura T, Nawata H. Dihydrotestosterone suppresses foam cell formation and attenuates atherosclerosis development. Endocrinology. 2010 Jul;151(7):3307-16. doi: 10.1210/en.2009-1268. Epub 2010 Apr 28. PMID 20427482
- [Background] Rettew JA, Huet-Hudson YM, Marriott I. Testosterone reduces macrophage expression in the mouse of toll-like receptor 4, a trigger for inflammation and innate immunity. Biol Reprod. 2008 Mar;78(3):432-7. doi: 10.1095/biolreprod.107.063545. Epub 2007 Nov 14. PMID 18003947
- [Background] Ribas V, Drew BG, Le JA, Soleymani T, Daraei P, Sitz D, Mohammad L, Henstridge DC, Febbraio MA, Hewitt SC, Korach KS, Bensinger SJ, Hevener AL. Myeloid-specific estrogen receptor alpha deficiency impairs metabolic homeostasis and accelerates atherosclerotic lesion development. Proc Natl Acad Sci U S A. 2011 Sep 27;108(39):16457-62. doi: 10.1073/pnas.1104533108. Epub 2011 Sep 7. PMID 21900603
- [Background] Kratz M, Purnell JQ, Breen PA, Thomas KK, Utzschneider KM, Carr DB, Kahn SE, Hughes JP, Rutledge EA, Van Yserloo B, Yukawa M, Weigle DS. Reduced adipogenic gene expression in thigh adipose tissue precedes human immunodeficiency virus-associated lipoatrophy. J Clin Endocrinol Metab. 2008 Mar;93(3):959-66. doi: 10.1210/jc.2007-0197. Epub 2007 Dec 18. PMID 18089690
- [Background] Herbst KL, Anawalt BD, Amory JK, Bremner WJ. Acyline: the first study in humans of a potent, new gonadotropin-releasing hormone antagonist. J Clin Endocrinol Metab. 2002 Jul;87(7):3215-20. doi: 10.1210/jcem.87.7.8675. PMID 12107227
- [Background] Herbst KL, Coviello AD, Page S, Amory JK, Anawalt BD, Bremner WJ. A single dose of the potent gonadotropin-releasing hormone antagonist acyline suppresses gonadotropins and testosterone for 2 weeks in healthy young men. J Clin Endocrinol Metab. 2004 Dec;89(12):5959-65. doi: 10.1210/jc.2003-032123. PMID 15579744
- [Background] Page ST, Herbst KL, Amory JK, Coviello AD, Anawalt BD, Matsumoto AM, Bremner WJ. Testosterone administration suppresses adiponectin levels in men. J Androl. 2005 Jan-Feb;26(1):85-92. PMID 15611571
- [Background] Bhasin S, Storer TW, Berman N, Callegari C, Clevenger B, Phillips J, Bunnell TJ, Tricker R, Shirazi A, Casaburi R. The effects of supraphysiologic doses of testosterone on muscle size and strength in normal men. N Engl J Med. 1996 Jul 4;335(1):1-7. doi: 10.1056/NEJM199607043350101. PMID 8637535
- [Background] Tricker R, Casaburi R, Storer TW, Clevenger B, Berman N, Shirazi A, Bhasin S. The effects of supraphysiological doses of testosterone on angry behavior in healthy eugonadal men--a clinical research center study. J Clin Endocrinol Metab. 1996 Oct;81(10):3754-8. doi: 10.1210/jcem.81.10.8855834.
- [Background] Bhasin S, Woodhouse L, Casaburi R, Singh AB, Mac RP, Lee M, Yarasheski KE, Sinha-Hikim I, Dzekov C, Dzekov J, Magliano L, Storer TW. Older men are as responsive as young men to the anabolic effects of graded doses of testosterone on the skeletal muscle. J Clin Endocrinol Metab. 2005 Feb;90(2):678-88. doi: 10.1210/jc.2004-1184. Epub 2004 Nov 23. PMID 15562020
- [Background] Cuzick J, DeCensi A, Arun B, Brown PH, Castiglione M, Dunn B, Forbes JF, Glaus A, Howell A, von Minckwitz G, Vogel V, Zwierzina H. Preventive therapy for breast cancer: a consensus statement. Lancet Oncol. 2011 May;12(5):496-503. doi: 10.1016/S1470-2045(11)70030-4. PMID 21441069
- [Background] Leder BZ, LeBlanc KM, Schoenfeld DA, Eastell R, Finkelstein JS. Differential effects of androgens and estrogens on bone turnover in normal men. J Clin Endocrinol Metab. 2003 Jan;88(1):204-10. doi: 10.1210/jc.2002-021036. PMID 12519853
- [Background] Belgorosky A, Guercio G, Pepe C, Saraco N, Rivarola MA. Genetic and clinical spectrum of aromatase deficiency in infancy, childhood and adolescence. Horm Res. 2009;72(6):321-30. doi: 10.1159/000249159. Epub 2009 Oct 21. PMID 19844120
- [Background] Campbell KL, Makar KW, Kratz M, Foster-Schubert KE, McTiernan A, Ulrich CM. A pilot study of sampling subcutaneous adipose tissue to examine biomarkers of cancer risk. Cancer Prev Res (Phila). 2009 Jan;2(1):37-42. doi: 10.1158/1940-6207.CAPR-08-0073. PMID 19139016
- [Background] Muniyappa R, Lee S, Chen H, Quon MJ. Current approaches for assessing insulin sensitivity and resistance in vivo: advantages, limitations, and appropriate usage. Am J Physiol Endocrinol Metab. 2008 Jan;294(1):E15-26. doi: 10.1152/ajpendo.00645.2007. Epub 2007 Oct 23. PMID 17957034
- [Background] Olefsky JM, Glass CK. Macrophages, inflammation, and insulin resistance. Annu Rev Physiol. 2010;72:219-46. doi: 10.1146/annurev-physiol-021909-135846. PMID 20148674
- [Derived] Rubinow KB, Vaisar T, Chao JH, Heinecke JW, Page ST. Sex steroids mediate discrete effects on HDL cholesterol efflux capacity and particle concentration in healthy men. J Clin Lipidol. 2018 Jul-Aug;12(4):1072-1082. doi: 10.1016/j.jacl.2018.04.013. Epub 2018 Apr 30. PMID 29793828
- [Derived] Chao J, Rubinow KB, Kratz M, Amory JK, Matsumoto AM, Page ST. Short-Term Estrogen Withdrawal Increases Adiposity in Healthy Men. J Clin Endocrinol Metab. 2016 Oct;101(10):3724-3731. doi: 10.1210/jc.2016-1482. Epub 2016 Aug 2. PMID 27482750

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 06/01/13-11/30/2014 Location: University/Medical Center Flyers, newspaper ads, online postings
Pre-assignment Details: 116 subjects were screened, 63 subjects didn't meet study inclusion/exclusion criteria or they withdrew consent prior to group assignment, and 3 subjects withdrew prior to the baseline visit.
Groups:
- Acyline & Placebo Gel & Placebo Pill: Acyline (300mcg/kg at Day 0 & week 2, by injections) + placebo transdermal gel + placebo aromatase inhibitor daily for 4 weeks
  Acyline: 300 mcg/mL administered subcutaneously (at Day 0, Week 2)
  Placebo gel (for Testosterone 1.62% gel): placebo gel manufactured to mimic Testosterone 1.62% gel
  Placebo pill (for Letrozole): Oral placebo aromatase inhibitor to mimic Letrozole 5mg/d
- Acyline & Testosterone Gel 1.25g/d & Placebo Pill: Acyline (300mcg/kg at Day 0 & week 2, by injections) + Testosterone 1.62% gel (1.25g) daily + placebo aromatase inhibitor pill daily for 4 weeks
  Acyline: 300 mcg/mL administered subcutaneously (at Day 0, Week 2)
  Testosterone 1.62% gel: Transdermal Testosterone Gel (either 3.75g or 5g/d) for 4 weeks
  Placebo pill (for Letrozole): Oral placebo aromatase inhibitor to mimic Letrozole 5mg/d
- Acyline & Testosterone Gel 5g/d & Placebo Pill: Acyline (300mcg/kg every 2 weeks, by injections) + Testosterone 1.62% gel (5g) daily + placebo aromatase inhibitor pill daily for 4 weeks
  Acyline: 300 mcg/mL administered subcutaneously (at Day 0, Week 2)
  Testosterone 1.62% gel: Transdermal Testosterone Gel (either 3.75g or 5g/d) for 4 weeks
  Placebo pill (for Letrozole): Oral placebo aromatase inhibitor to mimic Letrozole 5mg/d
- Acyline & Testosterone Gel & Letrozole: Acyline (300mcg/kg at Day 0 & week 2, by injections) + Testosterone transdermal 1.62% gel (5g) daily + letrozole (5mg) aromatase inhibitor pill daily for 4 weeks
  Acyline: 300 mcg/mL administered subcutaneously (at Day 0, Week 2)
  Testosterone 1.62% gel: Transdermal Testosterone Gel (either 3.75g or 5g/d) for 4 weeks
  Letrozole: Letrozole oral aromatase inhibitor 5mg daily for 4 weeks
Period: Overall Study
Arm/Group | Acyline & Placebo Gel & Placebo Pill | Acyline & Testosterone Gel 1.25g/d & Placebo Pill | Acyline & Testosterone Gel 5g/d & Placebo Pill | Acyline & Testosterone Gel & Letrozole
Started | 13 | 14 | 13 | 13
Completed | 12 | 13 | 12 | 13
Not Completed | 1 | 1 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — New Job | 0 | 1 | 0 | 0
Not completed — Weight Loss | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acyline & Placebo Gel & Placebo Pill | Acyline & Testosterone Gel 1.25g/d & Placebo Pill | Acyline & Testosterone Gel 5g/d & Placebo Pill | Acyline & Testosterone Gel & Letrozole | Total
Number analyzed (Participants) | 13 | 14 | 13 | 13 | 53
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 37 [27 to 51] | 35 [27 to 45] | 42 [31 to 51] | 34 [28 to 45] | 36 [29 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 13 | 14 | 13 | 13 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 9 | 11 | 11 | 13 | 44
  Unknown or Not Reported | 3 | 3 | 2 | 0 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 0 | 2 | 5
  White | 7 | 8 | 11 | 11 | 37
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 4 | 2 | 0 | 9
Region of Enrollment [Number; unit: participants]
  United States | 13 | 14 | 13 | 13 | 53
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 26 (4) | 26 (4) | 25 (2) | 25 (4) | 25 (3)
Weight [Mean (Standard Deviation); unit: kg] | 82 (14) | 81 (15) | 78 (8) | 82 (11) | 81 (12)
Fasting Glucose [Mean (Standard Deviation); unit: mg/dL] | 97 (6) | 97 (13) | 101 (7) | 98 (9) | 98 (9)
Percentage Body Fat [Mean (Standard Deviation); unit: %total body mass] | 28 (7) | 23 (6) | 24 (4) | 23 (7) | 24 (6)
Percentage Lean Mass [Mean (Standard Deviation); unit: %total body mass] | 68 (7) | 73 (5) | 72 (4) | 73 (7) | 72 (6)

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity Quantified by Matsuda Index
Description: Whole body insulin sensitivity as quantified by Matsuda Index at the end of the treatment period, calculated by the following equation: 10,000/square root of(FPG*FI)*(FPG+PG30*2+PG60*2+PG90*2+PG120)/8*(FPI+PI30*2+PI60*2+PI90*2+PI)/8). FPG=fasting plasma glucose level; FPI=fasting plasma insulin level; PG30,60,90, and 120=plasma glucose levels sampled at 30,60,90, and 120 minutes after oral glucose load; PI30,60,90, and 120=plasma insulin levels sampled at 30,60,90, and 120 minutes after the oral glucose load
Time Frame: 4 weeks
Population: Of the 53 subjects who attended the baseline study visit, 2 withdrew from the study and 1 was discontinued due to a protocol violation. 50 subjects completed the week 10 study visit. Of these, 5 subjects were excluded from the final analyses; 1 was found to have undiagnosed diabetes, and 4 subjects were excluded due to study drug non-adherence.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Acyline & Placebo Gel & Placebo Pill | Acyline & Testosterone Gel 1.25g/d & Placebo Pill | Acyline & Testosterone Gel 5g/d & Placebo Pill | Acyline & Testosterone Gel & Letrozole
Number analyzed (Participants) | 10 | 11 | 11 | 13
units on a scale | 5.0 [3.9 to 6.3] | 9.4 [4.5 to 14.0] | 7.2 [4.6 to 15.0] | 7.3 [5.9 to 10.0]
Statistical Analysis 1: Comparison: Acyline & Placebo Gel & Placebo Pill vs Acyline & Testosterone Gel 1.25g/d & Placebo Pill vs Acyline & Testosterone Gel 5g/d & Placebo Pill vs Acyline & Testosterone Gel & Letrozole; Test type: Superiority or Other; p = 0.164, RM-ANOVA — The a prior threshold for statistical significance was p<0.05

2. Secondary Outcome: Changes in Body Composition
Description: Fat mass and lean mass were measured by dual energy X-ray absorptiometry (DEXA) at baseline and at the end of the 4 week treatment period
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Acyline & Placebo Gel & Placebo Pill | Acyline & Testosterone Gel 1.25g/d & Placebo Pill | Acyline & Testosterone Gel 5g/d & Placebo Pill | Acyline & Testosterone Gel & Letrozole
Number analyzed (Participants) | 10 | 11 | 11 | 13
kg
  Change in fat mass | 1.1 (0.8) | 0.7 (0.5) | -0.4 (1.0) | 0.5 (0.8)
  Change in lean mass | -1.2 (1.0) | -1.4 (1.5) | 0.0 (1.0) | -0.3 (1.3)
Statistical Analysis 1: Comparison: Acyline & Placebo Gel & Placebo Pill vs Acyline & Testosterone Gel 1.25g/d & Placebo Pill vs Acyline & Testosterone Gel 5g/d & Placebo Pill vs Acyline & Testosterone Gel & Letrozole; Time-by-group interaction for fat mass; Test type: Superiority or Other; p = 0.003, RM-ANOVA
Statistical Analysis 2: Comparison: Acyline & Placebo Gel & Placebo Pill vs Acyline & Testosterone Gel 1.25g/d & Placebo Pill vs Acyline & Testosterone Gel 5g/d & Placebo Pill vs Acyline & Testosterone Gel & Letrozole; Test type: Superiority or Other; p = 0.03, RM-ANOVA — Time-by-group interaction for lean mass

3. Secondary Outcome: Changes in Adipose Tissue Gene Expression
Description: We examined whether differences in lipoprotein lipase expression would be evident across study treatment groups. RNA was isolated from whole adipose tissue gene expression, and complementary DNA (cDNA) was synthesized from 1.5 ug of RNA per sample. Gene expression was measured by polymerase chain reaction (PCR) using predesigned TaqMan® Gene Expression Assays. Standard curves were included on each plate, so Ct values were converted to copy numbers of the target gene. Expression values were normalized to the geometric mean of the housekeeping genes phosphoglycerate kinase and 18s.
Time Frame: 4 weeks
Population: Subjects were included who had adipose tissue samples available from both baseline and week 4 (end-of-treatment) visits.
Measure: Mean (Standard Deviation); unit: gene copy number per ng RNA
Groups:
- Acyline + Placebo Gel + Placebo Pills: Acyline (300 mg/kg, subcutaneous injection at weeks 0, 2) + placebo gel + oral placebo pills daily. This treatment regimen resulted in medical castration.
- Acyline + Testosterone Gel (1.25g/d) + Placebo Pills: Acyline (300 mcg/kg, subcutaneous injection at weeks 0, 2) + testosterone gel administered daily + daily placebo pills. This group was intended to have low-normal levels of serum testosterone and estradiol.
- Acyline + Testosterone Gel (5g/d) + Placebo Pills: Acyline (300 mcg/kg, subcutaneous injection at weeks 0, 2) + testosterone gel administered daily + daily placebo pills. This group was intended to have normal, physiologic levels of serum testosterone and estradiol.
- Acyline + Testosterone Gel (5g/d) + Letrozole: Acyline (300 mcg/kg, subcutaneous injection at weeks 0, 2) + testosterone gel administered daily + daily letrozole (pills). This group was intended to have normal levels of serum testosterone with selective estrogen deficiency.
Arm/Group | Acyline + Placebo Gel + Placebo Pills | Acyline + Testosterone Gel (1.25g/d) + Placebo Pills | Acyline + Testosterone Gel (5g/d) + Placebo Pills | Acyline + Testosterone Gel (5g/d) + Letrozole
Number analyzed (Participants) | 10 | 11 | 11 | 13
gene copy number per ng RNA | 7493 (1293) | 8224 (3485) | 7885 (2736) | 8320 (3133)
Statistical Analysis 1: Comparison: Acyline + Placebo Gel + Placebo Pills; The null hypothesis was that short-term testosterone deprivation would not affect lipoprotein lipase expression in adipose tissue. Repeated measures ANOVA was used to determine if a time-by-group effect was apparent for lipoprotein lipase expression; Test type: Other; p > 0.1, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse events were recorded through study completion, and subjects who experienced adverse events during the study were followed for up to 6 months after study participation ended.
Description: There were numerous, mild complications reported for the fat biopsy procedure such as bleeding, bruising, hematomas, tenderness, redness etc which are not listed. A frequency threshold of >15% was used for reported events.
Arm/Group | Acyline & Placebo Gel & Placebo Pill | Acyline & Testosterone Gel 1.25g/d & Placebo Pill | Acyline & Testosterone Gel 5g/d & Placebo Pill | Acyline & Testosterone Gel & Letrozole
Serious Adverse Events (participants affected / at risk) | 2/13 | 1/14 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 9/13 | 9/14 | 7/13 | 10/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acyline & Placebo Gel & Placebo Pill (N=13) | Acyline & Testosterone Gel 1.25g/d & Placebo Pill (N=14) | Acyline & Testosterone Gel 5g/d & Placebo Pill (N=13) | Acyline & Testosterone Gel & Letrozole (N=13)
Cardiac Arrthymia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abnormal Liver enzyme (AST & ALT) levels (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Elevated PSA level (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acyline & Placebo Gel & Placebo Pill (N=13) | Acyline & Testosterone Gel 1.25g/d & Placebo Pill (N=14) | Acyline & Testosterone Gel 5g/d & Placebo Pill (N=13) | Acyline & Testosterone Gel & Letrozole (N=13)
Hot Flashes (Endocrine disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Low libido (Endocrine disorders) | 4 (4) | 4 (4) | 0 (0) | 5 (5)
Erectile Dysfunction (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Low Energy (General disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Irritability (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Decreased testes size (Endocrine disorders) | 4 (4) | 2 (2) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No